CLINICAL TRIAL: NCT05707416
Title: Effect of Low Level Laser Therapy on Root Resorption During Orthodontic Intrusion of Maxillary Incisors: A Comparative Clinical Study
Brief Title: Effect of Low Level Laser Therapy on Root Resorption During Orthodontic Intrusion of Maxillary Incisors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Youssri Mahmoud Ahmed Saleh, doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 796/2193
Record Dates: First submitted 2022-11-22; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Root Resorption of Maxillary Incisors
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Will includes 9 patients who will receive intrusive arche after leveling and alignment assisted with laser with wavelength 635 nm, 6.5J/cm2,The laser will be applied to 4 points of application for each tooth two labial and two palatal started immediately after first intrusive wire then at days 3,7,14 and then every 15 day until achievement of the study objectives
  Interventions: Device: gallium aluminum arsenide (Ga-Al-As) semiconductor diode laser (SMARTTM PRO, LASOTRONIX, Poland)
- Control group (Active Comparator): Will includes 9 patients who will receive intrusive arches after leveling and alignment without laser application
  Interventions: Other: group B

INTERVENTIONS:
Device: gallium aluminum arsenide (Ga-Al-As) semiconductor diode laser (SMARTTM PRO, LASOTRONIX, Poland) — The laser will be applied to 4 points of application for each tooth two labial and two palatal started immediately after first intrusive wire then at days 3,7,14 and then every 15 day until achievement of the study objectives
  Arms: Experimental group
Other: group B — Will includes 9 patients who will receive intrusive arches after leveling and alignment without laser application
  Arms: Control group

SUMMARY:
The present study will be directed to evaluate the effect of low-level laser therapy on root resorption during orthodontic intrusion of upper incisors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age range between 12-16 years.

  * Overbite > 40% indicated for maxillary intrusion.
  * Mild to moderate crowding of upper incisors.
  * All permanent teeth erupted (excluding 3rd molars).
  * No previous orthodontic treatment.
  * Good oral hygiene with no previous periodontal surgery

Exclusion Criteria:

* Transverse and/or vertical skeletal dysplasia or craniofacial malformation.

  * Retained primary or missing permanent teeth in the maxillary anterior area, and any kind of tooth/root shape anomaly.
  * Patients with root resorption, impacted canines, or dental anomalies.
  * Poor oral hygiene
  * Present or history of periodontal diseases.
  * Systemic diseases or regular use of medications that could interfere with orthodontic tooth movement.
  * History of trauma affecting the maxillary incisors.
  * Endodontically treated upper anterior teeth.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
linear amount of root resorption | change in linear root resorption at 4 months
  cone beam computed linear measurements
volumetric amount of root resorption | change in volumetric root resorption at 4 months
  cone beam computed volumetric measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar Univertsity, Naşr, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goel P, Tandon R, Agrawal KK. A comparative study of different intrusion methods and their effect on maxillary incisors. J Oral Biol Craniofac Res. 2014 Sep-Dec;4(3):186-91. doi: 10.1016/j.jobcr.2014.11.007. Epub 2014 Dec 6. PMID 25737942